CLINICAL TRIAL: NCT02775851
Title: A Phase II and Pilot Trial of PD-1 Blockade With Pembrolizumab (MK-3475) in Patients With Resectable or Unresectable Desmoplastic Melanoma (DM)
Brief Title: Pembrolizumab in Treating Patients With Desmoplastic Melanoma That Can or Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-00666; NCI-2016-00666 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1512; S1512 (Other: SWOG); S1512 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Results first posted 2024-04-23 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Desmoplastic Melanoma
MeSH Terms: interventions — Biopsy; Specimen Handling; pembrolizumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (pembrolizumab, surgery) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles. Patients with potentially resectable disease undergo surgery. Patients with tumor progression and unresectable disease may receive one additional cycle of pembrolizumab. Patients undergo CT scan and may undergo PET and MRI throughout the study. Patients also undergo blood sample collection at screening and tumor biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Elastography; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Procedure: Therapeutic Conventional Surgery
- Cohort B (pembrolizumab) (Experimental): Patients with unresectable disease receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 34 cycles in the absence of disease progression or toxicity. Patients undergo CT scan and may undergo PET and MRI throughout the study. Patients also undergo blood sample collection at screening and tumor biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Elastography — Undergo MRI
  Other Names: MRE
  Arms: Cohort A (pembrolizumab, surgery)
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection

SUMMARY:
This pilot phase II trial studies how well pembrolizumab works in treating patients with desmoplastic melanoma (DM) that can be removed by surgery (resectable) or cannot be removed by surgery (unresectable). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the pathologic complete response rate (pCR) in patients with resectable desmoplastic melanoma treated with neoadjuvant pembrolizumab (MK-3475). (Cohort A) II. To evaluate the complete response rate (confirmed and unconfirmed) in patients with unresectable desmoplastic melanoma treated with pembrolizumab (MK-3475). (Cohort B)

SECONDARY OBJECTIVES:

I. To estimate the 9 week response rate (RR) (unconfirmed complete and partial responses) among patients with measurable disease. (Cohort A) II. To estimate the median overall survival (OS). (Cohort A) III. To evaluate safety and tolerability of pembrolizumab (MK-3475) in the neoadjuvant setting. (Cohort A) IV. To estimate the median progression-free survival (PFS). (Cohort B) V. To estimate the median overall survival (OS). (Cohort B) VI. To evaluate safety and tolerability of pembrolizumab (MK-3475) in this setting. (Cohort B)

OTHER OBJECTIVES:

I. To evaluate the hypothesis that higher mutational load in the patient derived baseline tumor biopsy samples is associated with higher pathologic complete response (pCR).

II. To evaluate T cell infiltration into the tumors and circulating tumor deoxyribonucleic acid (DNA) profile from blood samples in DM patients and correlate with response to programmed cell death protein 1 (PD-1) blockade.

III. To evaluate the clonality of tumor infiltrating T cells in DM patients and correlate with response to PD-1 blockade.

IV. To evaluate adaptive immune resistant mechanism in DM tumors.

OUTLINE: Patients are enrolled to 1 of 2 cohorts.

COHORT A: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles. Patients with potentially resectable disease undergo surgery. Patients with tumor progression and unresectable disease may receive one additional cycle of pembrolizumab.

COHORT B: Patients with unresectable disease receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 34 cycles in the absence of disease progression or toxicity.

Patients undergo computed tomography (CT) scan and may undergo position emission tomography (PET) and magnetic resonance imaging (MRI) throughout the study. Patients also undergo blood sample collection at screening and tumor biopsy throughout the study.

After completion of study treatment, patients are followed up at 6 weeks after the last dose, then every 12 weeks to the end of the first year, then every 6 months to the end of the fifth year after registration. After progression, patients are followed every 6 months for up to 2 years from the date of registration, then annually thereafter until 5 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* COHORT A: Patients must have histologically or cytologically confirmed primary desmoplastic melanoma that is deemed resectable; the decision to perform surgery on patients must be based on good clinical judgment; eligible patients for surgical resection must have disease that, in the judgment of the surgeon, is deemed completely resectable resulting in free surgical margins; patients must have residual disease after initial biopsy which can be measurable or non-measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; residual disease can either be confirmed with fine-needle aspiration (FNA) or if measurable disease is present, no FNA needs to be obtained OR
* COHORT B: Patients must have histologically or cytologically confirmed primary desmoplastic melanoma that is unresectable; patients in Cohort B must have measurable disease per RECIST 1.1
* Contrast-enhanced computed tomography (CT) scans of the chest, abdomen and pelvis are required; a whole body positron emission tomography (PET)/CT scan with diagnostic quality images and intravenous iodinated contrast may be used in lieu of a contrast enhanced CT of the chest, abdomen and pelvis; imaging of the head and neck is required only if the patient has a head/neck primary; contrast may be omitted if the treating investigator believes that exposure to contrast poses an excessive risk to the patient; if skin lesions are being followed as measurable disease, photograph with a ruler included and physician measurements, must be kept in the patient's chart as source documentation; all measurable lesions must be assessed within 28 days prior to registration; tests to assess non-measurable disease must be performed within 42 days prior to registration; all disease must be assessed and documented on the baseline tumor assessment form (RECIST 1.1)
* Patients must not have known brain metastases unless brain metastases have been treated and patient is asymptomatic with no residual neurological dysfunction and has not received enzyme-reducing anti-epileptic drugs or corticosteroids for at least 14 days prior to registration
* Patients must not have received prior systemic treatment for this melanoma
* Patients must not be planning to receive concomitant other biologic therapy, hormonal therapy, other chemotherapy, anti-cancer surgery or other anti-cancer therapy while on this protocol
* Patients must not have received radiation therapy, non-cytotoxic agents or investigational agents or systemic corticosteroids within 14 days prior to registration
* Patients may have received prior surgery; all adverse events associated with prior surgery must have resolved to =< grade 1 (per Common Terminology Criteria for Adverse Events [CTCAE] 4.0) prior to registration
* Patients must be >= 18 years of age
* Absolute neutrophil count (ANC) >= 1,500/mcl (obtained within 28 days prior to registration)
* Platelets >= 50,000/mcl (obtained within 28 days prior to registration)
* Hemoglobin >= 8 g/dL (obtained within 28 days prior to registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (or =< 3.0 x IULN with Gilbert's syndrome) (obtained within 28 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x IULN (or < 5 x IULN for patients with known liver metastases) (obtained within 28 days prior to registration)
* Patients must have lactate dehydrogenase (LDH) performed within 28 days prior to registration
* Patients must have Zubrod performance status =< 2
* Patients must not have history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Patients must not have an active infection requiring systemic therapy
* Patients must not have active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients must not have received live vaccines within 42 days prior to registration; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine; seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Patients known to be human immunodeficiency virus (HIV) positive prior to registration are eligible if they meet the following criteria within 30 days prior to registration: stable and adequate CD4 counts (>= 350 mm^3), and serum HIV viral load of < 25,000 IU/ml; patients must be on a stable anti-viral therapy
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated in situ cancer, adequately treated stage I or II cancer (including multiple primary melanomas) from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years
* Women of childbearing potential must have a negative urine or serum pregnancy test within 28 days prior to registration; women/men of reproductive potential must have agreed to use an effective contraceptive method for the course of the study through 120 days after the last dose of study medication; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy, or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures; patients must not be pregnant or nursing due to unknown teratogenic side effects
* Patients must have specimens available and institutions must be planning to submit for centralized pathology review and for integrated translational medicine objectives
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process, the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2026-05-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kari L Kendra, Principal Investigator — SWOG Cancer Research Network
Locations (281):
- United States (281):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope Upland, Upland, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Low Country Cancer Care, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Allegiance Health, Jackson, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Kendra KL, Bellasea SL, Eroglu Z, Hu-Lieskovan S, Campbell KM, Carson WE 3rd, Wada DA, Plaza JA, In GK, Ikeguchi A, Hyngstrom J, Brohl AS, Chmielowski B, Khushalani NI, Markowitz J, Monroe M, Contreras CM, Bowles T, Norman K, Medina E, Gonzalez CR, Baselga-Carretero I, Garcilazo IP, Vega-Crespo A, Chen JM, Deen NNA, Patel SP, Grossmann KF, Sondak VK, Sharon E, Moon J, Wu MC, Ribas A. Neoadjuvant PD-1 blockade in surgically resectable desmoplastic melanoma: cohort A of the phase 2 SWOG S1512 trial. Nat Cancer. 2026 Jan 29. doi: 10.1038/s43018-025-01113-y. Online ahead of print. PMID 41611998
- [Derived] Kendra KL, Bellasea SL, Eroglu Z, Hu-Lieskovan S, Campbell KM, Carson WE 3rd, Wada DA, Plaza JA, Sosman JA, In GK, Ikeguchi A, Hyngstrom J, Brohl AS, Khushalani NI, Markowitz J, Negrea G, Kasbari S, Doolittle GC, Swami U, Roberts T, Mathew BN, Medina E, Baselga-Carretero I, Gonzalez CR, Garcilazo IP, Vega-Crespo A, Chen JM, Naser Al-Deen N, Patel SP, Sharon E, Moon J, Wu MC, Ribas A. Anti-PD-1 therapy in unresectable desmoplastic melanoma: the phase 2 SWOG S1512 trial. Nat Med. 2025 Nov;31(11):3668-3674. doi: 10.1038/s41591-025-03875-5. Epub 2025 Aug 14. PMID 40813711

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 57 participants were enrolled, but one participant from Cohort A withdrew consent prior to receiving protocol treatment and is not analyzable.
Groups:
- Cohort A: Resectable - Pembrolizumab, Surgery: Resectable patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles. Patients with potentially resectable disease undergo surgery. Patients with tumor progression and unresectable disease may receive one additional cycle of pembrolizumab.
- Cohort B: Unresectable - Pembrolizumab: Unresectable patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 34 cycles in the absence of disease progression or toxicity.
Period: Overall Study
Arm/Group | Cohort A: Resectable - Pembrolizumab, Surgery | Cohort B: Unresectable - Pembrolizumab
Started | 30 | 27
Completed | 28 | 5
Not Completed | 2 | 22
Not completed — Adverse Event | 1 | 10
Not completed — Refusal Unrelated to Adverse Event | 0 | 1
Not completed — Progression/Relapse | 0 | 4
Not completed — Other - Not Protocol Specified | 0 | 7
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Resectable - Pembrolizumab, Surgery | Cohort B: Unresectable - Pembrolizumab | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Customized [Median (Full Range); unit: years]
  Age | 74.7 [37.3 to 91.1] | 75.2 [58.7 to 89.6] | 74.9 [37.3 to 91.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 22 | 25 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 28 | 27 | 55
  Race: Unknown | 1 | 0 | 1
Performance Status [Count of Participants; unit: Participants] — Zubrod Performance Status ranges from 0-4 w/ higher scores reflecting greater disability.
  0. Fully active, able to carry on all pre-disease performance w/o restriction
  1. Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature, e.g., light housework, office work
  2. Ambulatory & capable of self-care but unable to carry out any work activities; up & about >50% of waking hrs
  3. Capable of limited self-care, confined to bed or chair >50% of waking hrs
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair
  Participants
    0 | 22 | 19 | 41
    1 | 7 | 8 | 15
T Stage [Count of Participants; unit: Participants] — T category (primary tumor) criteria per the American Joint Committee on Cancer (AJCC) melanoma staging system (7th edition). TX means primary tumor cannot be assessed. T0 is no evidence of primary tumor. Tis is melanoma in situ. T1a is melanomas <= 1.0mm in thickness without ulceration and mitosis <1/mm^2. T1b is <=1.0mm with ulceration or mitosis >=1/mm^2. T2a is 1.01-2.0mm without ulceration. T2b is 1.01-2.0mm with ulceration. T3a is 2.01-4.0mm without ulceration. T3b is 2.01-4.0mm with ulceration. T4a is >4.0mm in thickness without ulceration. T4b is melanomas >4.0mm with ulceration.
  Participants
    Tis | 0 | 1 | 1
    T0 | 0 | 2 | 2
    T1a | 1 | 1 | 2
    T1b | 2 | 0 | 2
    T2a | 6 | 1 | 7
    T2b | 1 | 1 | 2
    T3a | 7 | 4 | 11
    T3b | 1 | 2 | 3
    T4a | 8 | 8 | 16
    T4b | 2 | 5 | 7
    Tx | 1 | 0 | 1
    Unknown | 0 | 2 | 2
N Stage [Count of Participants; unit: Participants] — N category (Regional Lymph Nodes) criteria per American Joint Committee on Cancer (AJCC) melanoma staging system (7th edition). NX mean regional nodes cannot be assessed. N0 = no regional metastases (mets) detected. N1a = 1 regional lymph node (LN) metastasis with micrometastasis. N1b = 1 regional LN metastasis with macrometastasis. N2a = 2-3 regional LN mets with micrometastasis. N2b = 2-3 regional LN mets with macrometastasis. N2c = In transit met(s)/satellite(s) without metastatic LNs. N3 is >=4 regional LN mets; or matted nodes; or in transit met(s)/satellite(s) with metastatic LN(s).
  Participants
    N0 | 24 | 12 | 36
    N1b | 2 | 2 | 4
    N2a | 0 | 1 | 1
    N2b | 0 | 2 | 2
    N2c | 3 | 1 | 4
    N3 | 0 | 2 | 2
    NX | 0 | 4 | 4
    Unknown | 0 | 3 | 3
M Stage [Count of Participants; unit: Participants] — M category (Distant Metastasis) criteria per American Joint Committee on Cancer (AJCC) melanoma staging system (7th edition). M0 is no detectable evidence of distant metastases. M1a is metastases to skin, subcutaneous or distant lymph nodes and normal serum LDH. M1b is metastases to lung and normal serum LDH. M1c is metastases to all other visceral sites and normal serum LDH or distant metastases to any site combined with an elevated serum LDH.
  Participants
    M0 | 29 | 8 | 37
    M1a | 0 | 1 | 1
    M1b | 0 | 11 | 11
    M1c | 0 | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate (Cohort A)
Description: Pathologic complete response is defined as no evidence of viable tumor cells on complete pathological evaluation of the surgical specimen per institutional standard of care.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Resectable - Pembrolizumab, Surgery
Number analyzed (Participants) | 29
percentage of participants | 55 [36 to 74]
Statistical Analysis 1: Comparison: Cohort A: Resectable - Pembrolizumab, Surgery; We assumed a null pCR rate of 5% and powered the study assuming an alternative hypothesis of 25%. This single stage design had an alpha of 3.4% (i.e. probability of declaring the regimen warrants further study when the true CR is 5%) and a power of 90% (probability of declaring the regimen warrants further study when the true pCR is 25%) with 25 eligible participants; Test type: Superiority; p < 0.001, One-sided Exact Binomial

2. Primary Outcome: Complete Response (CR) Rate (Cohort B)
Description: Complete response (per RECIST 1.1) defined as: disappearance of all target and non-target lesions no new lesions, no disease related symptoms, and any lymph nodes must have reduction in short axis to < 1.0 cm.
Time Frame: Up to 5 years
Population: All eligible and analyzable participants with measurable disease at baseline (n=27).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B: Unresectable - Pembrolizumab
Number analyzed (Participants) | 27
percentage of participants | 37 [19 to 58]
Statistical Analysis 1: Comparison: Cohort B: Unresectable - Pembrolizumab; We assumed a null CR rate of 5% and powered the study assuming an alternative hypothesis of 20%. This single stage design had an alpha of 8.5% (i.e. probability of declaring the regimen warrants further study when the true CR is 5%) and a power of 82% (probability of declaring the regimen warrants further study when the true CR is 20%) with 21 eligible participants; Test type: Superiority; p < 0.001, One-sided Exact Binomial

3. Secondary Outcome: 9 Week Response Rate (Cohort A)
Description: Unconfirmed complete (CR) and partial responses (PR) at end of neoadjuvant treatment assessment among patients with measurable disease. CR and PR per response evaluation criteria in solid tumors (RECIST v1.1): CR is complete disappearance of all target and non-target lesions, no new lesions, no disease related symptoms, and lymph nodes must have reduction in short axis to <1.0cm. PR is greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions, no unequivocal progression of non-measurable disease, and no new lesions. Overall response = CR + PR.
Time Frame: Up to 3 months
Population: All eligible and analyzable participants with measurable disease at baseline (n=26).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Resectable - Pembrolizumab, Surgery
Number analyzed (Participants) | 26
percentage of participants | 46 [27 to 67]

4. Secondary Outcome: Overall Survival (Cohort A and B)
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Resectable - Pembrolizumab, Surgery | Cohort B: Unresectable - Pembrolizumab
Number analyzed (Participants) | 29 | 27
months | NA [37.0 to NA] — There was insufficient follow-up data to estimate. | 50.6 [42.4 to NA] — There was insufficient follow-up data to estimate.

5. Secondary Outcome: Progression Free Survival (Cohort B)
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive without report of progression are censored at date of last contact. Progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST v1.1), as 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline, as well as an absolute increase of at least 0.5 cm, unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided), appearance of any new lesion/site, or death due to disease without prior documentation of progression and without symptomatic deterioration
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort B: Unresectable - Pembrolizumab
Number analyzed (Participants) | 27
months | 49.2 [33.3 to NA] — There was insufficient follow-up data to estimate.

6. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. CTCAE Version 4.0 was used for all AE reporting.
Time Frame: Duration of treatment and follow-up until death or 5 years post registration.
Population: Participants who were eligible and received at least one dose of protocol treatment. 29 participants were evaluable or AEs in Cohort A and 27 were evaluable or AEs in Cohort B.
Measure: Number; unit: Participants
Groups:
- Cohort A: MK-3475 (Pembrolizumab): Resectable patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles. Patients with potentially resectable disease undergo surgery. Patients with tumor progression and unresectable disease may receive one additional cycle of pembrolizumab.
- Cohort B: MK-3475 (Pembrolizumab): Unresectable patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 34 cycles in the absence of disease progression or toxicity.
Arm/Group | Cohort A: MK-3475 (Pembrolizumab) | Cohort B: MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 29 | 27
Participants
  Abdominal pain | 0 | 1
  Adrenal insufficiency | 0 | 1
  Back pain | 0 | 1
  CPK increased | 0 | 1
  Colitis | 1 | 2
  Diarrhea | 0 | 2
  Dyspnea | 0 | 1
  Hypokalemia | 0 | 1
  Hypoxia | 0 | 1
  Immune system disorders - Other, specify | 0 | 1
  Lipase increased | 0 | 1
  Lung infection | 0 | 1
  Mucositis oral | 1 | 0
  Musculoskeletal and connective tiss disorder - Other | 0 | 1
  Myositis | 0 | 1
  Pancreatitis | 0 | 2
  Rash maculo-papular | 0 | 2
  Sepsis | 0 | 1
  Skin and subcutaneous tissue disorders - Other | 0 | 1
  Upper gastrointestinal hemorrhage | 0 | 1

7. Other Pre Specified Outcome: Baseline Mutational Load (Cohort A and B)
Description: Will assess the association between per megabase mutation rate and pCR or CR status.
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in T-cell Infiltration (Cohort A and B)
Description: Will compare change in CD8 expression following treatment between responders and non-responders.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: ctDNA Fraction
Description: Will assess the association between response and ctDNA fraction.
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Clonality of Tumor Infiltrating T Cells (Cohort A and B)
Description: Will compare change from baseline in TCR clonality metric between responders and non-responders.
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Adaptive Immune Resistant Mechanism (Cohort A and B)
Description: Will compare change in PD-L1 expression between responders and non-responders.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 5 years post registration.
Description: CTCAE version 4.0 was used for toxicity SAEs reporting. There were 29 participants in Cohort A that were assessed for AEs and 27 participants Cohort B that were assessed for AEs.
Arm/Group | Cohort A: MK-3475 (Pembrolizumab) | Cohort B: MK-3475 (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 5/29 | 10/27
Serious Adverse Events (participants affected / at risk) | 1/29 | 14/27
Other Adverse Events (participants affected / at risk) | 23/29 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: MK-3475 (Pembrolizumab) (N=29) | Cohort B: MK-3475 (Pembrolizumab) (N=27)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Immune system disorders-Other (Immune system disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
CPK increased (Investigations) | 0 | 1
Cardiac troponin I increased (Investigations) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: MK-3475 (Pembrolizumab) (N=29) | Cohort B: MK-3475 (Pembrolizumab) (N=27)
Anemia (Blood and lymphatic system disorders) | 4 | 11
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 4
Blurred vision (Eye disorders) | 0 | 2
Cataract (Eye disorders) | 0 | 2
Eye disorders-Other (Eye disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 4 | 6
Diarrhea (Gastrointestinal disorders) | 8 | 9
Dysphagia (Gastrointestinal disorders) | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 5
Vomiting (Gastrointestinal disorders) | 1 | 2
Edema limbs (General disorders) | 0 | 3
Facial pain (General disorders) | 1 | 2
Fatigue (General disorders) | 16 | 20
Flu like symptoms (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 3
Pain (General disorders) | 4 | 6
Skin infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 4
Alkaline phosphatase increased (Investigations) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 6
Blood bilirubin increased (Investigations) | 0 | 2
Creatinine increased (Investigations) | 1 | 5
Lymphocyte count decreased (Investigations) | 2 | 7
Platelet count decreased (Investigations) | 1 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 5
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 5
Hypernatremia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 4
Hypokalemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 3 | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Dizziness (Nervous system disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 5 | 5
Memory impairment (Nervous system disorders) | 1 | 3
Paresthesia (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 5
Depression (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 6
Hematuria (Renal and urinary disorders) | 1 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 8
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 8
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 2 | 5
Hypotension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02775851/Prot_SAP_000.pdf